CLINICAL TRIAL: NCT00734097
Title: An Open Label, Multicentre Study of Nexium (Esomeprazole) 40 mg Once Daily in Subjects With Symptoms of Gastroesophageal Reflux Disease (GORD) After Treatment With a Full Dose of Proton Pump Inhibitor (PPI)
Brief Title: A Study of Nexium (Esomeprazole) 40 mg Once Daily in Subjects With Symptoms of Gastroesophageal Reflux Disease (GORD) After Treatment With a Full Dose of Proton Pump Inhibitor (PPI)
Acronym: NEON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9612L00116; NEON
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Results first posted 2012-10-10 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-08

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: heartburn; reflux; proton; pump; inhibitor
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Esomeprazole; Restraint, Physical; Pregnancy Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nexium 40 mgs (Experimental)
  Interventions: Drug: Esomeprazole 40 mg; Procedure: Physical Exam; Other: Quality of Life Questionnaires; Procedure: pregnancy test, if applicable

INTERVENTIONS:
Drug: Esomeprazole 40 mg — Once a day
  Other Names: Nexium
Procedure: Physical Exam — every visit
Other: Quality of Life Questionnaires — every visit
Procedure: pregnancy test, if applicable — as needed

SUMMARY:
The purpose of this study is to assess how patients with gastro-oesophageal reflux disease (heartburn) who are currently receiving treatment with a proton pump inhibitor but are still experiencing symptoms will benefit from a change in treatment.

ELIGIBILITY:
Inclusion Criteria:

* Persisting symptoms of GORD despite previous treatment with a full dose proton pump inhibitor
* informed consent
* over 18 years of age

Exclusion Criteria:

* Current course of Proton Pump inhibitor treatment for more than 8 weeks prior to enrolment in the study
* More than 1 other course of PPI treatment in the previous 12 month
* previous use of esomeprazole
* presence of alarm symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Research Site, Buenos Aires, Argentina
- Chile (3):
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- Colombia (3):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Medellín
- Venezuela (3):
  - Research Site, Barquisimeto
  - Research Site, Caracas
  - Research Site, San Cristóbal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with persisting symptoms of Gastroesophageal Reflux Disease (GORD) despite previous treatment with a full dose proton pump inhibitor were enrolled across the Argentina (6 sites), Chile (3 sites) Colombia (9 sites) and Venezuela (2 sites).
Pre-assignment Details: All participants received 8-weeks open label esomeprazole treatment.
Groups:
- Esomeprazole 40mg, Daily: Open-label daily esomeprazole 40 mg, daily for 8 weeks
Period: Screening
Arm/Group | Esomeprazole 40mg, Daily
Started | 337
Completed | 317 (20 participants were screening failure.)
Not Completed | 20
Not completed — Protocol Violation | 12
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 2
Not completed — Unconfirmed pregnancy | 1
Period: Open Label
Arm/Group | Esomeprazole 40mg, Daily
Started | 317 (Full analysis performed in 311)
Safety Analysis | 317
Full Analysis | 311
Per Protocol | 301
Completed | 301 (16 patients discontinued after randomization)
Not Completed | 16
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 5
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Arm/Group | Esomeprazole 40mg, Daily
Number analyzed (Participants) | 311
Age Continuous [Mean (Standard Deviation); unit: Years] — Age at study entry
  Years | 42.7 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender
  Participants
    Female | 212
    Male | 99

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Days With Heartburn From Baseline to 8 Weeks of Treatment
Description: Reported frequency of days with heartburn at week 8 - reported frequency of days with heartburn at baseline
Time Frame: At Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Days per week with symptoms
Arm/Group | Esomeprazole 40mg, Daily
Number analyzed (Participants) | 311
Days per week with symptoms | -3.44 (2.35)

2. Secondary Outcome: Change in Frequency of Days With Heartburn From Baseline to 4 Weeks of Treatment
Description: Reported frequency of days with heartburn at week 4 - reported frequency of days with heartburn at baseline.
Time Frame: At Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: Days per week with symptoms
Arm/Group | Esomeprazole 40mg, Daily
Number analyzed (Participants) | 311
Days per week with symptoms | -3.08 (2.32)

3. Secondary Outcome: Change in Severity of Heartburn From Baseline to 8 Weeks of Treatment
Description: Reported severity of heartburn at week 8 on RDQ - reported severity of heartburn at baseline on RDQ RDQ: Reflux Disease Questionnaire - by AstraZeneca LLP, 2000, values from "None" to "Severe".
  Four dimensions are defined for the RDQ - heartburn, regurgitation, GORD dimension and dyspepsia: stomach. Scores for each dimension are range from 0 to 5 for frequency (not present to daily) and/or severity (not present to severe).
Time Frame: At Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Units of scale
Arm/Group | Esomeprazole 40mg, Daily
Number analyzed (Participants) | 311
Units of scale | -1.56 (1.01)

4. Secondary Outcome: Change in Severity of Heartburn From Baseline to 4 Weeks of Treatment
Description: Reported severity of heartburn at week 4 on RDQ - reported severity of heartburn at baseline on RDQ (RDQ: Reflux Disease Questionnaire - by AstraZeneca LLP, 2000, values from "None" to "Severe".
  Four dimensions are defined for the RDQ - heartburn, regurgitation, GORD dimension and dyspepsia: stomach. Scores for each dimension are range from 0 to 5 for frequency (not present to daily) and/or severity (not present to severe).
Time Frame: At Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Esomeprazole 40mg, Daily
Number analyzed (Participants) | 311
Units on scale | -1.34 (1.03)

5. Secondary Outcome: Change in Frequency of Days With Acid Regurgitation From Baseline to 4 Weeks of Treatment.
Description: Reported frequency of days with Acid regurgitation at week 4 - reported frequency of days with acid regurgitation at baseline.
  Four dimensions are defined for the Reflux Disease Questionnaire (RDQ) - heartburn, regurgitation, GORD dimension and dyspepsia: stomach. Scores for each dimension are range from 0 to 5 for frequency (not present to daily) and/or severity (not present to severe).
Time Frame: At Baseline and 4 weeks.
Measure: Mean (Standard Deviation); unit: Days per week with symptoms
Arm/Group | Esomeprazole 40mg, Daily
Number analyzed (Participants) | 311
Days per week with symptoms | -2.95 (2.42)

6. Secondary Outcome: Change in Frequency of Days With Acid Regurgitation From Baseline to 8 Weeks of Treatment.
Description: Reported frequency of days with Acid regurgitation at week 8 - reported frequency of days with acid regurgitation at baseline.
  Four dimensions are defined for the Reflux Disease Questionnaire (RDQ) - heartburn, regurgitation, GORD dimension and dyspepsia: stomach. Scores for each dimension are range from 0 to 5 for frequency (not present to daily) and/or severity (not present to severe).
Time Frame: At Baseline and 8 weeks.
Measure: Mean (Standard Deviation); unit: Days per week with symptoms
Arm/Group | Esomeprazole 40mg, Daily
Number analyzed (Participants) | 311
Days per week with symptoms | -3.28 (2.51)

7. Secondary Outcome: Change in Frequency of Epigastric Pain After 4 Weeks of Treatment
Description: Reported frequency of days with Epigastric Pain at week 4 - reported frequency of days with Epigastric Pain at baseline.
  Four dimensions are defined for the Reflux Disease Questionnaire (RDQ) - heartburn, regurgitation, GORD dimension and dyspepsia: stomach. Scores for each dimension are range from 0 to 5 for frequency (not present to daily) and/or severity (not present to severe).
Time Frame: At Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: Days per week with pain
Arm/Group | Esomeprazole 40mg, Daily
Number analyzed (Participants) | 311
Days per week with pain | -2.77 (2.5)

8. Secondary Outcome: Change in Frequency of Epigastric Pain After 8 Weeks of Treatment
Description: Reported frequency of days with Epigastric Pain at week 8 - reported frequency of days with Epigastric Pain at baseline.
  Four dimensions are defined for the Reflux Disease Questionnaire (RDQ) - heartburn, regurgitation, GORD dimension and dyspepsia: stomach. Scores for each dimension were range from 0 to 5 for frequency (not present to daily) and severity (not present to severe).
Time Frame: At Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Days per week with pain
Arm/Group | Esomeprazole 40mg, Daily
Number analyzed (Participants) | 311
Days per week with pain | -3.16 (2.52)

9. Secondary Outcome: Change in Severity of Epigastric Pain After 8 Weeks of Treatment
Description: Reported severity of epigastric pain at week 8 on RDQ - reported severity of epigastric pain at baseline on RDQ (RDQ: Reflux Disease Questionnaire - by AstraZeneca LLP, 2000, values from "None" to "Severe".
  Four dimensions are defined for the RDQ - heartburn, regurgitation, GORD dimension and dyspepsia: stomach. Scores for each dimension are range from 0 to 5 for frequency (not present to daily) and/or severity (not present to severe).
Time Frame: At Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Units of scale
Arm/Group | Esomeprazole 40mg, Daily
Number analyzed (Participants) | 311
Units of scale | -1.34 (1.1)

10. Secondary Outcome: Change in Severity of Epigastric Pain After 4 Weeks of Treatment
Description: Reported severity of epigastric pain at week 4 on RDQ - reported severity of epigastric pain at baseline on RDQ (RDQ: Reflux Disease Questionnaire - by AstraZeneca LLP, 2000, values from "None" to "Severe".
  Four dimensions are defined for the RDQ - heartburn, regurgitation, GORD dimension and dyspepsia: stomach. Scores for each dimension are range from 0 to 5 for frequency (not present to daily) and/or severity (not present to severe).
Time Frame: At Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: Units of scale
Arm/Group | Esomeprazole 40mg, Daily
Number analyzed (Participants) | 311
Units of scale | -1.17 (1.1)

11. Secondary Outcome: Change in Severity of Acid Regurgitation After 8 Weeks of Treatment
Description: Reported severity of acid regurgitation at week 8 on RDQ - reported severity of acid regurgitation at baseline on RDQ (RDQ: Reflux Disease Questionnaire - by AstraZeneca LLP, 2000, values from "None" to "Severe".
  Four dimensions are defined for the RDQ - heartburn, regurgitation, GORD dimension and dyspepsia: stomach. Scores for each dimension are range from 0 to 5 for frequency (not present to daily) and/or severity (not present to severe).
Time Frame: At Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Units of scale
Arm/Group | Esomeprazole 40mg, Daily
Number analyzed (Participants) | 311
Units of scale | -1.51 (1.09)

12. Secondary Outcome: Change in Severity of Acid Regurgitation After 4 Weeks of Treatment
Description: Reported severity of acid regurgitation at week 4 on RDQ - reported severity of acid regurgitation at baseline on RDQ (RDQ: Reflux Disease Questionnaire - by AstraZeneca LLP, 2000, values from "None" to "Severe".
  Four dimensions are defined for the RDQ - heartburn, regurgitation, GORD dimension and dyspepsia: stomach. Scores for each dimension are range from 0 to 5 for frequency (not present to daily) and/or severity (not present to severe).
Time Frame: At Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: Units of scale
Arm/Group | Esomeprazole 40mg, Daily
Number analyzed (Participants) | 311
Units of scale | -1.31 (1.06)

ADVERSE EVENTS:
Arm/Group | Esomeprazole 40mg, Daily
Serious Adverse Events (participants affected / at risk) | 4/317
Other Adverse Events (participants affected / at risk) | 16/317
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 40mg, Daily (N=317)
Dizziness / Hypotension / Tachycardia (Cardiac disorders) | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Uterine Leiomyoma (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 40mg, Daily (N=317)
Headache (Nervous system disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less